CLINICAL TRIAL: NCT04549948
Title: Curve of Spee: Speed of Leveling Using Different Orthodontic Archwire Size and Material - A Randomized Clinical Trial
Brief Title: Curve of Spee: Speed of Leveling Using Different Orthodontic Archwires
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Elham Abu Alhaija, Professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 436/2018
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Orthodontic Treatment
Keywords: root resorption; pain; pulpal blood flow
MeSH Terms: conditions — Root Resorption; Pain

STUDY DESIGN:
Intervention Model Description: Leveling of the curve of Spee
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient was blinded to the intervention used. However, it was not possible to blind the clinician during treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.017X0.025 Stainless Steel Archwire (Experimental): Leveling of COS using 0.017X0.025 Stainless Steel (SS) Archwire A reverse COS using 0.017X0.025 SS was used to correct the excessive COS in the lower arch.
  Interventions: Procedure: 0.017X0.025 Stainless steel
- 0.019X0.025 Stainless Steel Archwire (Experimental): A reverse COS using 0.019X0.025 SS was used to correct the excessive COS in the lower arch.
  Interventions: Procedure: 0.019X0.025 Stainless steel
- 0.021X0.025 TMA archwire (Experimental): A reverse COS using 0.021X0.025 TMA archwire was used to correct the excessive COS in the lower arch.
  Interventions: Procedure: 0.021X0.025 B-Titanium archwire

INTERVENTIONS:
Procedure: 0.017X0.025 Stainless steel — Leveling curve of Sppe using 0.017X0.025 SS archwire
  Arms: 0.017X0.025 Stainless Steel Archwire
Procedure: 0.019X0.025 Stainless steel — Leveling curve of Sppe using 0.019X0.025 Stainless steel archwire
  Arms: 0.019X0.025 Stainless Steel Archwire
Procedure: 0.021X0.025 B-Titanium archwire — Leveling curve of Sppe using 0.019X0.025 B-Titanium archwire
  Arms: 0.021X0.025 TMA archwire

SUMMARY:
The objectives if this study was to evaluate the efficacy of 3 different rectangular archwires in the correction of the curve of Spee (COS), to record the time needed to level excessive COS in the mandibular arch using the 3 archwire sizes, to investigate the changes in intercanine and intermolar widths and arch length during leveling, to measure the arterio-posterior and vertical movement for the lower incisors and lower molars, to record pulpal blood flow and to detect the root resorption in the lower anterior teeth associated with leveling excessive COS using the 3 different archwires.

DETAILED DESCRIPTION:
Fifty one subjects with an excessive COS were included in this study. The subjects will be randomly divided into three groups; Group one (17 patients): leveling of COS using 0.017X0.025-inch stainless steel archwire. Group two (17 patients): leveling of COS using 0.019X0.025-inch stainless steel archwire. Group three (17 patients): leveling of COS using 0.021X0.025-inch Titanium molybdenum archwire.

In the three groups, a 5mm depth reverse COS will be inserted. Records consisted of lateral cephalograms (pre-treatment, at T0 and post-treatment), peri-apical radiographs (at T0 and at T5), study casts (pre-treatment and at each time point during the tudy). Patients will be followed up on monthly visits without removing leveling archwires where alginate impressions were taken for the lower arch. Pain scores during the first week of leveling will be recorded using visual analogue scale (VAS).The amount of COS correction in mm, changes in intercanine in mm, intermolar and arch length in mm, pain scores and lower incisors root resorptions in mm will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years and ≤ 30 years
* Overbite covering more than half of the lower incisor height
* Curve of Spee ≥ 4 millimeters
* Mild crowding in lower arch where non-extraction treatment is indicated.
* Normally inclined or retroclined lower incisors
* Averaged or reduced lower vertical height
* Good oral hygiene and healthy periodontium
* All permanent teeth are present except for the third molars

Exclusion Criteria:

* Severe crowding in lower arch where extraction treatment is indicated.
* Missing permanent molars or Premolars
* Poor oral hygiene and Periodontal disease
* Systemic health problems and medications were taken
* History of previous orthodontic treatment
* Smoking

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Curve of Spee depth changes during leveling | 4 to 6 months
  The change in Curve of Spee in millimetres

SECONDARY OUTCOMES:
Pain perception | one week
  A10-point visual analogue scale of 10 cm length where 0 indicate no pain and 10 indicate intolerable pain
Root Resorption | 6 months
  change in root length in millimeters
Pulpal blood flow | one month
  Change in blood flow using laser flowmetry

CONTACTS AND LOCATIONS:
Overall Officials: Elham S A Abu Alhaija, PhD, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ba-Hattab R, Abu Alhaija ES, Nasrawi YH, Taha N, Daher H, Daher S. Leveling the curve of Spee using different sized archwires: a randomized clinical trial of blood flow changes. Clin Oral Investig. 2023 Jun;27(6):2943-2955. doi: 10.1007/s00784-023-04894-7. Epub 2023 Feb 11. PMID 36773128